CLINICAL TRIAL: NCT05008692
Title: Measuring Cardiopulmonary Fitness in Ambulatory Heart Failure Patients Through the Use of Apple Watch Features
Brief Title: Apple-CPET Ted Rogers Understanding Exacerbations of Heart Failure
Acronym: TRUE-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Apple Inc. (Industry)
Responsible Party: Principal Investigator, Heather Ross, Chief Division of Cardiology, University Health Network, Toronto
Other Study IDs: 20-5205
Record Dates: First submitted 2021-07-24; First posted 2021-08-17 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure; Heart Failure, Systolic; Heart Failure, Diastolic; Heart Transplantation; Heart Failure，Congestive
Keywords: Wearable; Apple Watch; Cardiopulmonary Exercise Test; 6MWT; Biomarker; peak VO2; Patient Reported Outcomes; QOL
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart Failure (HF) is a complex disease associated with the highest burden of cost to the healthcare system. The cardiopulmonary exercise test (CPET) is instrumental in determining the prognosis of patients with HF. This study will evaluate whether aggregate biometric data from the Apple Watch combined with demographic, cardiac, and biomarker testing can improve our ability to predict heart failure outcomes among a diverse ambulatory HF population

DETAILED DESCRIPTION:
Heart Failure (HF) has a prevalence of 3.5% suggesting that over one million Canadians are affected by this disease, and more than 50,000 are newly diagnosed each year. This complex disease is associated with the highest burden of cost to the healthcare system, attributable to hospitalizations, missed work, medications, and health care services

Traditionally, clinicians have relied on static snapshots of patients to determine clinical status and estimate prognosis. More advanced cardiac centers rely on cardiopulmonary exercise testing (CPET), where patients are further stratified based on validated exercise parameters. CPET remains underutilized and resource-intensive. It requires expensive equipment, proficient personnel, and clinicians with specialized training. Thus, there is an unmet need for a more widely available, accessible, and longitudinal assessment of clinical status to better monitor and prognosticate patients outside of the ambulatory setting. Wearable devices such as the Apple Watch hold great promise in this regard, as they provide near-continuous monitoring of biometric data. By combining biometric data with demographic, cardiac, and biomarker testing, the investigators will significantly improve our ability to predict heart failure outcomes such as early warning of decompensation, clinical deterioration (symptoms and brain natriuretic peptide (BNP) as a surrogate), hospitalization, mortality (using the Seattle Heart Failure Model (SHFM) as a surrogate), and/or need for advanced heart failure therapies.

Our study has 5 research questions based on 2 primary outcomes and 3 secondary outcomes in clinically diverse adult ambulatory heart failure patients :

Primary Research Question:

1. Can biometric data obtained from the Apple Watch be used to estimate cardiorespiratory fitness, as assessed by CPET?
2. Does the 'predicted' Apple 6 MW estimate correlate with formal 6 MWT?

   Secondary Research Questions:
3. Is there a relationship between novel biosensors, including oxygen saturation, and markers of poor prognosis specifically as defined by the SHFM, BNP, Quality of life (QOL) indicators, and CPET parameters?
4. Can surrogates of cardiorespiratory fitness obtained from the Apple Watch, including novel biosensors, predict acute decompensation of heart failure as defined rapid clinic visits, need for IV diuretics, ED visits, heart failure hospitalization and unscheduled health care encounters during the 3-month follow-up?
5. Can biometric data be used to improve a risk prediction model that can distinguish between patients at high versus low risk of all-cause hospitalization (primary outcome), all-cause mortality (secondary outcome), and a composite outcome of all-cause mortality, need for ventricular assist device, or heart transplantation (secondary composite outcome) over a 2 year period?

ELIGIBILITY:
Inclusion Criteria:

* broad age range (> 17 years of age)
* diverse races/ethnicities,
* equal female and male representation,
* NYHA functional class I-IV, heart failure with reduced and preserved ejection fraction

Exclusion

- Physical disability that prevents exercise testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>17 years of age), ambulatory heart failure patients currently followed by the University Health Network.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Apple Watch metrics prediction of CPET parameters | 3 months
  Measure predictive power of Apple Watch metrics such as heart rate against CPET parameters such as peak VO2
6 minute walk test | 3 months
  Correlation of Apple 6MW estimate with measured 6MWT

SECONDARY OUTCOMES:
Apple Watch sensors and markers of poor prognosis | 3 months
  Correlation between novel biosensors, including oxygen saturation, and markers of poor prognosis specifically as defined by the Seattle Heart Failure Model (SHFM), BNP, Quality of life (QOL) and CPET parameters
Apple Watch Sensors and unscheduled visits | 3 months
  Identify whether Apple Watch sensors including estimated peak VO2 predict a composite outcome of unscheduled visits (including: rapid clinic visits, need for IV diuretics, ED visit and HF hospitalization)
Biomarkers and digital signatures as a predictor of composite rehospitalisation, advanced therapies and mortality | 2 years
  Identify novel biomarkers (eg. ST2, cell-free DNA, peripheral markers of the microbiome) collected by the biobank and digital signatures assessed by the Apple Watch (eg. behaviors, exercise, medication adherence) that predict a composite outcome of mortality, advanced heart failure therapies and hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Ross, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Moayedi Y, Foroutan F, Gao Y, Kim B, De Luca E, Brum M, Brahmbhatt DH, Duhamel J, Simard A, McIntosh C, Ross HJ. Developments in Digital Wearable in Heart Failure and the Rationale for the Design of TRUE-HF (Ted Rogers Understanding of Exacerbations in Heart Failure) Apple CPET Study. Circ Heart Fail. 2025 Jun;18(6):e012204. doi: 10.1161/CIRCHEARTFAILURE.124.012204. Epub 2025 May 9. PMID 40340421